CLINICAL TRIAL: NCT02871570
Title: A Phase 1, Non-randomized, Open-label, Parallel-group Single-dose Study To Evaluate The Pharmacokinetics, Safety, And Tolerability Of Intravenous Rivipansel (Pf-06460031) In Subjects With Moderate Hepatic Impairment And In Healthy Subjects With Normal Hepatic Function
Brief Title: A Study to Evaluate the Effect of IV Doses of Rivipansel in Subjects With Moderate Hepatic Impairment and in Healthy Subjects With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlycoMimetics Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: B5201006
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Results first posted 2018-11-28 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Moderate Hepatic Impairment; Normal Hepatic Function
Keywords: Hepatic Impairment; Rivipansel
MeSH Terms: interventions — rivipansel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moderate Hepatic Impairment (Experimental): A single dose of IV Rivipansel over 20 minutes
  Interventions: Drug: Rivipansel
- Normal Hepatic Function (Experimental): A single dose of IV Rivipansel over 20 minutes
  Interventions: Drug: Rivipansel

INTERVENTIONS:
Drug: Rivipansel — A single dose of IV Rivipansel over 20 minutes
  Other Names: GMI-1070

SUMMARY:
The purpose of this study is to determine the effect of hepatic impairment on rivipansel PK and safety.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of non-childbearing potential or male subjects

  * Body Mass Index (BMI) of 17.5 to 40.0 kg/m2
  * Normal Hepatic function for the healthy subjects
  * Stable Hepatic Impairment for the subjects with moderate hepatic impairment

Exclusion Criteria:

* Treatment with an investigational drug within 30 days of the dose of study medication
* Pregnant females, breastfeeding female subjects and male subjects with partners currently pregnant
* Use of herbal supplements in the 28 days prior to the dose of study medication
* Blood donation (excluding plasma donation) of approximately 1 pint or more within 56 days prior to study medication
* A positive urine drug screen for illicit drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Orlando Clincial Research Center, Orlando, Florida, United States

REFERENCES:
- [Derived] Tammara BK, Ryan K, Plotka A, Shafer FE, Wei H, Readett D, Fang A, Korth-Bradley JM. Effect of Renal or Hepatic Impairment on the Pharmacokinetics, Safety, and Tolerability of Intravenous Rivipansel. Clin Pharmacol Drug Dev. 2020 Nov;9(8):918-928. doi: 10.1002/cpdd.842. Epub 2020 Jun 24. PMID 32579796

RESULTS

PARTICIPANT FLOW:
Groups:
- Moderate Hepatic Impairment Group: A single dose of rivipansel 840 mg was administered intravenously (IV) to a group of participants with moderate hepatic impairment.
- Normal Hepatic Function Group: A single dose of rivipansel 840 mg was administered intravenously (IV) to a group of participants with normal hepatic function.
Period: Overall Study
Arm/Group | Moderate Hepatic Impairment Group | Normal Hepatic Function Group
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who received study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Hepatic Impairment Group | Normal Hepatic Function Group | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.00 (3.85) | 58.75 (4.43) | 58.38 (4.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Post-baseline Clinically Significant Findings in Physical Examinations
Description: A full physical examination was performed for each participant, and it included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes and gastrointestinal, musculoskeletal, and neurological systems. Clinical significance of laboratory findings was determined by the investigator.
Time Frame: Day 5
Population: Safety analysis set included all participants who received study medication.
Measure: Number; unit: participants
Arm/Group | Moderate Hepatic Impairment Group | Normal Hepatic Function Group
Number analyzed (Participants) | 8 | 8
participants | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product or medical device, regardless of its causal relationship with study treatment. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; was life-threatening (immediate risk of death); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs were events between administration of study medication and up to follow-up visit (28-31 days after administration) that were absent before treatment or that worsened after treatment. AEs included both serious and non-serious AEs.
Time Frame: Day 1 to follow-up visit (28-31 days after administration of study medication on Day 1)
Population: Safety analysis set included all participants who received study medication.
Measure: Number; unit: participants
Arm/Group | Moderate Hepatic Impairment Group | Normal Hepatic Function Group
Number analyzed (Participants) | 8 | 8
participants
  AEs | 1 | 1
  SAEs | 0 | 0

3. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Pre-defined Summarization Criteria
Description: Maximum absolute values and increases from baseline were summarized for PR interval (time from the beginning of P wave to the start of QRS complex, corresponding to the end of atrial depolarization and onset of ventricular depolarization), QRS duration (time from Q wave to the end of S wave, corresponding to ventricle depolarization), and QTcF interval (time from the beginning of Q wave to the end of T wave corresponding to electrical systole corrected for heart rate using Fridericia's formula). Number of participants with ECG findings meeting the following criteria is presented: (1) PR interval >=300 msec; (2) QRS duration >=200 msec; (3) QTcF interval: 450 to <480 msec; (4) QTcF interval: 480 to <500 msec; (5) QTcF interval >=500 msec; (6) PR interval percent increase from baseline >=25/50 percent; (7) QRS duration percent increase from baseline >=50 percent; (8) QTcF interval increase from baseline: 30 to <60 msec; (9) QTcF interval increase from baseline >=60 msec.
Time Frame: Day 5
Population: Safety analysis set included all participants who received study medication.
Measure: Number; unit: participants
Arm/Group | Moderate Hepatic Impairment Group | Normal Hepatic Function Group
Number analyzed (Participants) | 8 | 8
participants
  PR interval >=300 msec | 0 | 0
  QRS duration >=200 msec | 0 | 0
  QTcF interval: 450 to <480 msec | 1 | 0
  QTcF interval: 480 to <500 msec | 0 | 0
  QTcF interval >=500 msec | 0 | 0
  PR interval increase from baseline >=25/50 percent | 0 | 0
  QRS duration increase from baseline >=50 percent | 0 | 0
  QTcF increase from baseline: 30 to <60 msec | 0 | 0
  QTcF interval increase from baseline >=60 msec | 0 | 0

4. Primary Outcome: Number of Participants With Vital Signs Data Meeting Pre-defined Summarization Criteria
Description: Absolute values and changes from baseline (increase and decrease) were summarized for supine diastolic blood pressure (DBP), supine systolic blood pressure (SBP), and supine pulse rate. Number of participants with vital signs findings meeting the following criteria is presented: (1) supine DBP <50 millimeters of mercury (mm Hg); (2) supine DBP >90 mm Hg; (3) supine SBP <90 mm Hg; (4) supine SBP >140 mm Hg (for normal hepatic function group); (5) supine SBP >160 mm Hg (for moderate hepatic impairment group); (6) supine pulse rate < 40 beats per minute (bpm); (7) supine pulse rate >120 bpm; (8) supine DBP increase from baseline >=20 mm Hg; (9) supine SBP increase from baseline >=30 mmHg; (10) supine DBP decrease from baseline >=20 mm Hg; (11) supine SBP decrease from baseline >=30 mm Hg.
Time Frame: Day 1 to Day 5
Population: Safety analysis set included all participants who received study medication.
Measure: Number; unit: participants
Arm/Group | Moderate Hepatic Impairment Group | Normal Hepatic Function Group
Number analyzed (Participants) | 8 | 8
participants
  supine DBP <50 mm Hg | 0 | 0
  supine DBP >90 mm Hg | 0 | 0
  supine SBP <90 mm Hg | 0 | 0
  supine SBP >140 mm Hg (normal function group): number analyzed (Participants) | 0 | 8
  supine SBP >140 mm Hg (normal function group) |  | 0
  supine SBP >160 mm Hg (moderate impairment group): number analyzed (Participants) | 8 | 0
  supine SBP >160 mm Hg (moderate impairment group) | 0 |
  supine pulse rate <40 bpm | 0 | 0
  supine pulse rate >120 bpm | 0 | 0
  supine DBP increase from baseline >=20 mm Hg | 1 | 0
  supine SBP increase from baseline >=30 mmHg | 1 | 0
  supine DBP decrease from baseline >=20 mm Hg | 0 | 0
  supine SBP decrease from baseline >=30 mm Hg | 0 | 0

5. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: Laboratory tests included: hematology (hemoglobin, hematocrit, red and white blood cell count, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes, prothrombin time/international normalized ratio), chemistry (blood urea nitrogen/urea and creatinine, fasting glucose, calcium, sodium, potassium, chloride, total carbon dioxide, aspartate and alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid, albumin, total protein), urinalysis (pH, qualitative glucose, protein, and blood, ketones, nitrites, leukocyte esterase, urobilinogen, urine bilirubin, and microscopy), and other tests (follicle stimulating hormone, urine drug test and serologic tests on human immunodeficiency virus-1 antibody, Hepatitis B surface antigen and hepatitis C antibody). Abnormality was determined by the investigator using widely accepted criteria in clinical practice.
Time Frame: Day 5
Population: Safety analysis set included all participants who received study medication.
Measure: Number; unit: participants
Arm/Group | Moderate Hepatic Impairment Group | Normal Hepatic Function Group
Number analyzed (Participants) | 8 | 8
participants | 7 | 0

6. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) of Rivipansel
Description: AUCinf was calculated as AUClast + (Clast*/kel), where Clast* was the predicted plasma concentration at the last quantifiable time point estimated from the log linear regression analysis, kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Pre-dose, 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post-dose on Day 1
Population: The pharmacokinetic (PK) parameter analysis population included all participants treated who had at least one of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/milliliter (hr*mcg/mL)
Arm/Group | Moderate Hepatic Impairment Group | Normal Hepatic Function Group
Number analyzed (Participants) | 8 | 8
hour*microgram/milliliter (hr*mcg/mL) | 599.7 (25) | 770.0 (14)
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment Group vs Normal Hepatic Function Group; Test type: Other; ratio = 0.7789, 90% CI 2-sided [0.6514 to 0.9313] — Moderate hepatic impairment group represents the numerator, and normal hepatic function group represents the denominator

7. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of Rivipansel
Description: Area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (AUClast) of rivipansel was determined using a linear/log trapezoidal method.
Time Frame: Pre-dose, 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post-dose on Day 1
Population: The PK parameter analysis population included all participants treated who had at least one of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*mcg/mL
Arm/Group | Moderate Hepatic Impairment Group | Normal Hepatic Function Group
Number analyzed (Participants) | 8 | 8
hr*mcg/mL | 593.8 (26) | 763.7 (14)
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment Group vs Normal Hepatic Function Group; Test type: Other; ratio = 0.7776, 90% CI 2-sided [0.6493 to 0.9311] — [estimate comment as in outcome 6, analysis 1]

8. Primary Outcome: Total Clearance From Plasma (CL) of Rivipansel
Description: CL of rivipansel was calculated as dose/AUCinf, where AUCinf referred to the area under the plasma concentration-time profile from time 0 extrapolated to the infinite time.
Time Frame: Pre-dose, 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post-dose on Day 1
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour
Arm/Group | Moderate Hepatic Impairment Group | Normal Hepatic Function Group
Number analyzed (Participants) | 8 | 8
liter/hour | 1.401 (26) | 1.091 (14)
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment Group vs Normal Hepatic Function Group; Test type: Other; ratio = 1.2844, 90% CI 2-sided [1.0732 to 1.5372] — [estimate comment as in outcome 6, analysis 1]

9. Secondary Outcome: Maximum Observed Concentration (Cmax) of Rivipansel
Time Frame: Pre-dose, 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post-dose on Day 1
Population: The PK concentration population included all participants treated who had at least 1 PK concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Moderate Hepatic Impairment Group | Normal Hepatic Function Group
Number analyzed (Participants) | 8 | 8
mcg/mL | 77.91 (38) | 98.06 (28)
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment Group vs Normal Hepatic Function Group; Test type: Other; ratio = 0.7945, 90% CI 2-sided [0.5955 to 1.0599] — [estimate comment as in outcome 6, analysis 1]

10. Secondary Outcome: Terminal Half-Life of Rivipansel
Description: Terminal half-life of rivipansel was calculated as loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve.
Time Frame: Pre-dose, 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post-dose on Day 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Moderate Hepatic Impairment Group | Normal Hepatic Function Group
Number analyzed (Participants) | 8 | 8
hours | 7.653 (0.964) | 7.805 (0.923)

11. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Rivipansel
Description: Vss of rivipansel was calculated as CL*MRT, where MRT was the mean residence time and CL was the clearance from plasma.
Time Frame: Pre-dose, 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post-dose on Day 1
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Moderate Hepatic Impairment Group | Normal Hepatic Function Group
Number analyzed (Participants) | 8 | 8
liters | 14.08 (29) | 11.20 (14)

12. Other Pre Specified Outcome: Time for Maximum Observed Concentration (Tmax) of Rivipansel
Time Frame: Pre-dose, 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post-dose on Day 1
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Moderate Hepatic Impairment Group | Normal Hepatic Function Group
Number analyzed (Participants) | 8 | 8
hours | 0.667 [0.667 to 3.33] | 0.667 [0.667 to 0.667]

ADVERSE EVENTS:
Time Frame: Day 1 to follow-up visit (28-31 days after administration of study medication on Day 1)
Arm/Group | Moderate Hepatic Impairment Group | Normal Hepatic Function Group
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Hepatic Impairment Group (N=8) | Normal Hepatic Function Group (N=8)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-06-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT02871570/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT02871570/SAP_001.pdf